CLINICAL TRIAL: NCT02639091
Title: An Open Label Phase Ib Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Maximum Tolerated Dose of Anetumab Ravtansine in Combination With Pemetrexed 500 mg/m2 and Cisplatin 75 mg/m2 in Subjects With Mesothelin-expressing Predominantly Epithelial Mesothelioma or Nonsquamous Non-small-cell Lung Cancer
Brief Title: Phase Ib Study of Anetumab Ravtansine in Combination With Pemetrexed and Cisplatin in Mesothelin-expressing Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17631; 2016-003988-18 (EudraCT Number)
Record Dates: First submitted 2015-11-30; First posted 2015-12-24 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Medical Oncology
Keywords: Phase 1; Solid tumors; Mesothelioma; Lung cancer; Pemetrexed; Cisplatin
MeSH Terms: conditions — Mesothelioma; Lung Neoplasms | interventions — anetumab ravtansine; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAY 94-9343 + Pemetrexed + Cisplatin (Experimental): Investigating the combination of anetumab ravtansine (BAY 94-9343) with Pemetrexed (500 mg/m2) and Cisplatin (75 mg/m2) in Part 1 (dose escalation cohorts) and Part 2 (two MTD expansion cohorts)
  Interventions: Drug: BAY 94-9343; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: BAY 94-9343 — In Part 1 of the study, anetumab ravtansine (BAY 94-9343) will be administered by 1-hour IV infusion with a starting dose of 5.5mg/kg(BW) on Day 1 of every treatment cycle (Q3W).
  In Part 2 of the study, anetumab ravtansine (BAY 94-9343) will be administered on Day 2 of Cycle 1 and then on Day 1 of Cycle 2 and all subsequent cycles (Q3W)
Drug: Pemetrexed — Administered at the dose of 500 mg/m2 body surface area (BSA) by 10-minute IV infusion on Day 1 of every treatment cycle (Q3W) in both parts of the study
Drug: Cisplatin — Administered at the dose of 75 mg/m2 (BSA) by 2-hour IV infusion on Day 1 of every treatment cycle (Q3W) in both parts of the study

SUMMARY:
Determine the safety, tolerability and maximum tolerated dose of anetumab ravtansine (BAY 94-9343) in combination with pemetrexed 500 mg/m2 and cisplatin 75 mg/m2 in subjects with mesothelin-expressing predominantly epithelial mesothelioma or nonsquamous non-small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be male or female, and must be aged =/>18 years on the date of signing the informed consent form.
* Subjects must have histologically confirmed, unresectable, locally advanced or metastatic pleural or peritoneal predominantly (>50% of tumor component) epithelial mesothelioma or nonsquamous non-small-cell lung cancer (NSCLC). Both chemotherapy-naive and previously treated subjects will be eligible; however, newly diagnosed NSCLC subjects eligible for FDA-approved therapies should have received the same before enrollment (e.g. subjects with epidermal growth factor receptor [EGFR]-mutated and anaplastic lymphoma kinase [ALK]-translocated NSCLC should have received FDA-approved targeted therapies).
* Subjects must have at least 1 measurable or evaluable tumor lesion according to RECIST 1.1 (for nonsquamous NSCLC) or mRECIST (for epithelial pleural mesothelioma). Subjects with resected primary tumors who have documented metastases are eligible.
* Subjects must have a life expectancy of at least 12 weeks.
* Subjects must have ECOG (Eastern Cooperative Oncology Group performance Status of 0 or 1
* Subjects must have adequate bone marrow, liver, kidney, and coagulation functions.

Exclusion Criteria:

* Subjects who have a previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study, or any previous cancer curatively treated >3 years before the start of study Treatment.
* Subjects who have a history or current evidence of bleeding disorder, i.e. any hemorrhage / bleeding event of CTCAE (Common Terminology Criteria for Adverse Events) Grade ≥2 within 4 weeks before the start of study Treatment.
* Subjects who have new or progressive brain or meningeal or spinal metastases.
* Subjects who have a history or current evidence of uncontrolled cardiovascular disease i.e. NYHA (New York Heart Association) Class III or IV.
* Subjects who have a history or current evidence of uncontrolled hypertension defined as systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg at screening despite optimal medical management.
* Subjects who have a history or current evidence of malignant biliary obstruction requiring biliary stent.
* Subjects who have had solid organ or bone marrow Transplantation.
* Subjects who have a history of hypersensitivity to any of the study drugs or their excipients, or a history of severe hypersensitivity to any other Antigen.
* Subjects who have a history of human immunodeficiency virus (HIV) infection or subjects who have an active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection requiring treatment.
* Subjects who have an active clinically serious infection of CTCAE Grade ≥2 or non-healing wound unrelated to the primary Tumor.
* Subjects who have received systemic cancer therapy, radiotherapy, investigational drug treatment outside of this study within 4 weeks before the start of study treatment, granulocyte colony stimulating factors, (G-CSF) or granulocyte macrophage-stimulating factors (GM-CSF), erythropoietin-stimulating agents within 3 weeks before the start of general screening, drugs with known renal toxicity and strong cytochrome P450 3A4 (CYP3A4) inhibitors or strong CYP3A4 inducers within 2 weeks before the treatment.
* Subjects who have started oral or parenteral anticoagulation therapy within 2 weeks before the start of anetumab ravtansine until end of treatment visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 2 years
  MTD is defined as the highest dose of oral anetumab ravtansine (BAY 94-9343) administered in combination with IV pemetrexed and cisplatin that can be given such that not more than 1 of 6 subjects at a given dose level experience a DLT (dose-limiting toxicity).
Number of subjects with adverse events and serious adverse events as a measure of safety and tolerability | Up to 2 years

SECONDARY OUTCOMES:
Plasma concentrations of anetumab ravtansine (BAY 94-9343), pemetrexed and cisplatin | - BAY 94-9343: C1D1,D2,D3,D8,D15, C2D1, C3D1,D2,D3,D8,D15, C4D1, C6D1 and subsequent cycles every 3rd cycle up to 2 years or until discontinuation of study treatment, whichever comes first - Pemetrexed: C1D1, D2, D3 - Cisplatin: C1D1, D2, D3
  C (treatment cycle), D (day); Each cycle is defined as a period of 21 days
Tumor response evaluation following mRECIST criteria to determine the number of patients with CR, PR, SD or PD | Baseline, every 8 weeks up to cycle 12; then every 12 weeks from cycle 13 up to 2 years, or until discontinuation of study treatment, whichever comes first
  CR (complete response); PR (partial response); SD (stable disease); PD (progressive disease); Each cycle is defined as a period of 21 days
Number of patients with a positive titer of anti-drug antibodies | Day1 of C1, C3, C6 and subsequent cycles every 3rd cycle up to 2 years or until discontinuation of study treatment, whichever comes first
  Each cycle is defined as a period of 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- United States (4):
  - Chicago, Illinois
  - Bethesda, Maryland
  - Detroit, Michigan
  - Charleston, South Carolina
- Milan, Lombardy, Italy